CLINICAL TRIAL: NCT01786850
Title: Magnetic Resonance-guided High-intensity Focused Ultrasound Treatment of Locally Advanced Pancreatic Cancer: Phase II Study for Pain Palliation and Local Tumor Control
Brief Title: Magnetic Resonance-guided High-intensity Focused Ultrasound Treatment of Locally Advanced Pancreatic Cancer
Status: Available | Type: Expanded Access
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Napoli, MD, PhD, University of Roma La Sapienza
Other Study IDs: Pancreafus-01
Record Dates: First submitted 2013-02-05; First posted 2013-02-08 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Pancreas; Cancer; Locally Advanced Pancreatic Cancer; Non-invasive Treatment
Keywords: Locally advanced Pancreatic Cancer; Noninvasive treatment; High Intensity focused ultrasound; Magnetic Resonance
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Procedure: Magnetic Resonance-guided High-intensity Focused Ultrasound (MRgFUS) — High intensity focused ultrasound (HIFU) is a non-invasive ablation technique under ultrasound (US) guidance for the treatment of solid tumors. Differently from other ablations, HIFU induces tissue necrosis through short (10-30s) and relatively low grade (60-80 C°) thermal stimulations. Clinical applications of HIFU include uterine fibroids, prostate, hepatic and breast cancer. Selected patients with pancreatic cancer have been treated with US-guided HIFU for both pain control and tumor debulking. The development of a MR guidance for HIFU (MRgFUS) enabled to perform real-time monitoring and precise control of beam direction, temperature changes and deposited thermal dose beyond the capability of conventional US guidance. This system has been approved for the treatment of uterine fibroids and bone metastases in the United States and European Union. As compared to conventional US-guided HIFU, MRgFUS could represent a more accurate ablation modality for unresectable pancreatic cancer.

SUMMARY:
Patients with unresectable pancreatic cancer in most of cases cannot benefit from percutaneous ablation modalities, due to high risk of procedure-related complications. Ultrasound-guided high intensity focused ultrasound (HIFU) ablation has been introduced as a feasible treatment option in these patients. However, in other anatomical regions US-guided HIFU has been replaced by the more accurate MR-guided focused ultrasound (MRgFUS) ablation, but the applicability of this latter technique to the treatment of pancreatic cancer is still unexplored. The aim of this study is to explore feasibility and clinical performance of MRgFUS ablation of unresectable pancreatic cancer. Two are the main end-points: Pain palliation and local tumor control.

As compared to conventional US-guided HIFU, MRgFUS could represent a more accurate, non-invasive ablation modality even for unresectable pancreatic cancer although, to date, no cases of pancreatic MRgFUS ablation have been reported.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven unresectable pancreatic adenocarcinoma;
* unable or not willing to undergo chemo-radiation therapy
* Celiac plexus alcoholization failed to control pain symptoms

Exclusion Criteria:

* contraindication to MR or general anesthesia

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: alessandro napoli, Principal Investigator — Sapienza University of Rome, Policlinico Umberto I Hospital; carlo catalano, Study Chair — Sapienza University of Rome, Policlinico Umberto I Hospital; michele anzidei, Study Director — Sapienza University of Rome, Policlinico Umberto I Hospital
Locations (1):
- Sapienza University of Rome, Policlinico Umberto I Hospital, Rome, Italy